CLINICAL TRIAL: NCT02197468
Title: Gut Microbiome Study in Preterm Infants - a Norwegian Multi Centre Study
Brief Title: Preterm Infant Gut (PINGU) - a Norwegian Multi Centre Study
Acronym: PINGU
Status: Completed | Type: Observational
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); Oslo University Hospital (Other); Ullevaal University Hospital (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014/930 (REK)
Record Dates: First submitted 2014-07-21; First posted 2014-07-22 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2016-06

CONDITIONS: Mixed Flora; Infection
Keywords: Gut microbiome; Necrotizing enterocolitis; Antibiotics
MeSH Terms: conditions — Infections; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Fecal samples for bacterial DNA analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Probiotics: Preterm infants given probiotics: GA 24-27 weeks/Birth weight < 1000 g
  Preterm infants not given probiotics: GA 28-31 weeks/Birth weight 1000-1500 g
  Full-term infants not given probiotics (control)

SUMMARY:
Necrotizing enterocolitis (NEC) is a leading cause of morbidity and mortality among infants in the neonatal intensive care unit (NICU). It has been postulated that abnormal colonization of the preterm gut, or an unfavorable balance between gut bacteria may contribute to the development of NEC.

Recent clinical randomized studies and meta-analysis have shown that proactive colonization of probiotic bacteria reduce the frequency of NEC. Based on this evidence, in April 2014 all Norwegian NICUs started routinely administration of probiotics to all extremely premature neonates susceptible to NEC (gestational age <28 weeks/birth weight <1000g).

The current project is investigating the gut microbiome in patients receiving probiotics and compare the the gut microbiome with moderate premature infants not receiving probiotics. In addition, we are including a control of healthy full-term infants.

Samples containing feces from participants will be analyzed by state of the art whole-genome sequencing techniques. Bacterial diversity will be analysed with bioinformatic tools.

Study hypotheses:

* Probiotics given to extremely preterm infants will change the biodiversity of the gut microflora.
* Antibiotics given to these patients may influence the gut microflora also in infants receiving probiotics. In particular use of vancomycin may change the gut flora.
* After cessation of probiotic prophylaxis the gut flora of infants receiving probiotics will gradually resemble the gut flora of infants not receiving probiotics.
* A cross-contamination of probiotic bacteria between patients treated with probiotics and patients not treated with antibiotics may occur.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) is a leading cause of morbidity and mortality among infants in the neonatal intensive care unit (NICU). Prematurity is the most important risk factor for NEC. The pathogenesis of NEC remains unclear, and prevention and treatment strategies are limited. It has been postulated that abnormal colonization of the preterm gut, or an unfavorable balance between gut bacteria, is significant in the pathogenesis of NEC.

Recent clinical randomized studies and meta-analysis have shown that proactive colonization of probiotic bacteria reduce the frequency of NEC. Based on this evidence, in April 2014 all Norwegian NICUs started routinely administration of probiotics to all extremely premature neonates susceptible to NEC (gestational age (GA) <28 weeks/birth birth weight (BW) <1000 g).

The current project is investigating the gut microbiome in patients receiving probiotics and compare the the gut microbiome with moderate premature infants not receiving probiotics. In addition, we are including a control of healthy full-term infants.

Samples containing feces from participants will be analyzed by state of the art whole-genome sequencing techniques. Bacterial diversity and taxonomy will be analysed using bioinformatic tools

Inclusion criteria:

* Preterm infants 24-27 weeks gestation/ birth weight < 1000 g receiving probiotics
* Preterm infants 28-31 weeks gestation/BW 1000-1500 g not receiving probiotics
* Healthy term infants

Exclusion criteria

* Preterm infants < 24 weeks gestation
* Preterm infants < 32 weeks with severe lethal complication/poor prognosis around 1 week of age
* Infants with severe congenital malformations

Fecal samples will be obtained:

* 1 week of age
* 4 weeks of age
* 4 months corrected age
* 12 months corrected age

Study hypotheses:

* Probiotics given to extremely preterm infants will change the biodiversity of the gut microflora.
* Antibiotics given to these patients may influence the gut microflora also in infants receiving probiotics. In particular use of vancomycin may change the gut flora.
* After cessation of probiotic prophylaxis the gut flora of infants receiving probiotics will gradually resemble the gut flora of infants not receiving probiotics.
* A cross-contamination of probiotic bacteria between patients treated with probiotics and patients not treated with antibiotics may occur.

This is an explorative study. No formal sample size assessment is possible. Sequencing costs will be substantial. We will limit the number of participants to 26 x 2 preterm infants and 10 control healthy infants.

Six Norwegian Neonatal Intensive care units wil participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with gestational age 24-27 weeks/birth weight < 1000 g, treated with probiotics (target number 26)
* Preterm infants with gestational age 29-31 weeks/birth weight 1000-1500 g, not treated with probiotics (target number 26)
* Term infants (target number 10)

Exclusion Criteria:

* Extremely preterm infants with gestational age below 24 weeks
* Preterm infants (24-31 weeks) with life threatening complications during 1 week of age
* Infants with congenital malformations

Ages: 1 Hour to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants hospitalized in 6 Norwegian NICUs; divided in one group extremely preterm infants receiving probiotics and one group moderate preterm infants not receiving antibiotics. A group of helathy infants from the post-natal ward will also be included
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
To assess gut microbiome composition (meta genome sequencing) of preterm infants receiving probiotics versus preterm infants not receiving probiotics | 4 time points: 7 days of age, 4 weeks of age, 4 months corrected age and 12 months corrected age
  Stools samples from preterm infants and term infants (control)

SECONDARY OUTCOMES:
Impact of antibiotic exposure on gut microbiome | 4 time points: 7 days of age, 4 weeks of age, 4 months corrected age and 12 months corrected age
  Stool samples from preterm and term infants

OTHER OUTCOMES:
Cross contamination of probiotic bacteria in a NICU | 7 days of age and 4 weeks of age
  Detection of probiotic bacterial microbiome profiles in children not receiving probiotics

CONTACTS AND LOCATIONS:
Overall Officials: Claus Klingenberg, MD.phD.Prof., Study Chair — University Hospital of North Norway; Eirin Esaiassen, MD, Principal Investigator — University Hospital of North-Noway
Locations (7):
- Norway (7):
  - Haukeland Universtiy Hospital, Bergen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevaal, Oslo
  - Ahus University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim University Hospital, Trondheim

REFERENCES:
- [Background] Berrington JE, Stewart CJ, Cummings SP, Embleton ND. The neonatal bowel microbiome in health and infection. Curr Opin Infect Dis. 2014 Jun;27(3):236-43. doi: 10.1097/QCO.0000000000000061. PMID 24751892
- [Background] Stewart CJ, Marrs EC, Magorrian S, Nelson A, Lanyon C, Perry JD, Embleton ND, Cummings SP, Berrington JE. The preterm gut microbiota: changes associated with necrotizing enterocolitis and infection. Acta Paediatr. 2012 Nov;101(11):1121-7. doi: 10.1111/j.1651-2227.2012.02801.x. Epub 2012 Aug 31. PMID 22845166
- [Derived] Esaiassen E, Hjerde E, Cavanagh JP, Pedersen T, Andresen JH, Rettedal SI, Stoen R, Nakstad B, Willassen NP, Klingenberg C. Effects of Probiotic Supplementation on the Gut Microbiota and Antibiotic Resistome Development in Preterm Infants. Front Pediatr. 2018 Nov 16;6:347. doi: 10.3389/fped.2018.00347. eCollection 2018. PMID 30505830
- Available data/document: Clinical Study Report — https://www.frontiersin.org/articles/10.3389/fped.2018.00347/full — Publication from this study